CLINICAL TRIAL: NCT04198571
Title: MULTINATIONAL Retrospective Chart Review Study to Assess the Characteristics, Treatment Outcomes and Resource Use Among Adult Patients Hospitalised for Community-Acquired Pneumonia (CAP) or Complicated Skin and Soft Tissue Infections (cSSTI) Treated With Zinforo (REGISTERED) (Ceftaroline Fosamil) in a Usual Care Setting
Brief Title: Retrospective Chart Review Study to Assess Characteristics, Treatment Outcomes and Resource Use of Adults Hospitalized for CAP and CSSTi Treated With Zinforo in Multiple Countries
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C2661041
Record Dates: First submitted 2019-11-05; First posted 2019-12-13 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-09

CONDITIONS: Community Acquired Pneumonia; Complicated Skin and Soft Tissue Infection
Keywords: Bacteria; Zinforo® (ceftaroline fosamil); CAP; cSSTi; Hospitalized; Infectious Disease; Antibiotic; Cephalosporin
MeSH Terms: conditions — Community-Acquired Pneumonia; Soft Tissue Infections; Communicable Diseases | interventions — Ceftaroline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Not Applicable for this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Zinforo Treated: Only those Adults treated with this treatment for CAP or cSSTi
  Interventions: Drug: Zinforo (ceftaroline fosamil)

INTERVENTIONS:
Drug: Zinforo (ceftaroline fosamil) — IV Solution
  Other Names: Teflaro

SUMMARY:
MULTINATIONAL Retrospective Chart Review Study to Assess the Characteristics, Treatment Outcomes and Resource Use Among Adult Patients Hospitalized for Community-Acquired Pneumonia (CAP) or Complicated Skin and Soft Tissue Infections (cSSTI) Treated with Zinforo® (ceftaroline fosamil) in a Usual Care Setting

DETAILED DESCRIPTION:
The overall study aim is to provide real world evidence (RWE) on the characteristics, clinical management, treatment outcomes and healthcare resource use of adult patients aged 18 years and older admitted to the hospital for CAP or cSSTI who received Zinforo® in a usual care setting in Europe and Latin America on or before 31-May-2019.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 years or older at admission date to the hospital;
2. Received four (4) or more consecutive IV doses of Zinforo® in usual care on or before 31-May-2019; and
3. Admitting diagnosis to the hospital was either CAP or cSSTI.

Exclusion criteria:

1. Patients who were participating in an interventional clinical trial during the same hospital admission in which Zinforo® was administered;
2. Patients whose hospital medical records are missing documentation of the diagnostic criteria for either cSSTI or CAP;
3. Patients whose hospital medical records are missing details of dosing with Zinforo®;
4. Patients whose hospital medical records are missing information on the success/failure of Zinforo® treatment and the reason why treatment was discontinued; and
5. Patients whose hospital medical records are missing discharge date and status information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is adult patients aged 18 years and older hospitalized for CAP or cSSTI who received intravenous (IV) Zinforo® treatment in a usual care setting in Europe and Latin America on or before 31-May-2019.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2020-05-17 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- Brazil (2):
  - Real Hospital Português de Beneficência, Recife, Pernambuco
  - Hospital Esperança, Recife
- Colombia (4):
  - Clínica Las Américas, Medellín, Antioquia
  - E.S.E. Hospital Universitario San Jorge de Pereira, Pereira, Risaralda Department
  - Fundación Valle del Lili, Cali, Valle del Cauca Department
  - Centro médico Imbanaco, Cali
- France (4):
  - CHU Francois Mitterrand, Dijon
  - CHU de Grenoble Alpes, Grenoble
  - Croix-Rousse hospital, Hospices Civils de Lyon, Lyon
  - CHU Nantes, Nantes
- Greece (5):
  - Attikon University General Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - General University Hospital of Larissa, Larissa
  - Patras University Medical School, Pátrai
  - AHEPA General University Hospital of Thessaloniki, Thessaloniki
- Italy (5):
  - Asst Spedali Civili Brescia and Universita Degli Studi di Brescia, Brescia, Other
  - AORN Ospedali dei Colli - Ospedale Monaldi, Napoli, Other
  - Azienda Ospedaliera Dei Colli, Napoli
  - Aou Citta Della Salute E Della Scienza Scdu Malattie Infettive 2, Turin
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC), Presidio Ospedaliero Universitario Santa, Udine
- Russia (2):
  - Republican Clinical Hospital named after G.G. Kuvatova, Ufa, Bashkortostan Republic
  - BUZ UR First Republican Clinical Hospital under the Ministry of Healthcare of Udmurt Republic UR, Izhevsk, Udmurtiya Republic
- Spain (4):
  - Hospital Clínic, Barcelona
  - Hospital Universitario Valle de Hebrón, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Ferry T, Gogos C, Soriano A, Blasi F, Ansari W, Kantecki M, Schweikert B, Luna G, Bassetti M. Real-World Use and Treatment Outcomes of Ceftaroline Fosamil in Patients with Complicated Skin and Soft Tissue Infection: A Multinational Retrospective Study. Infect Drug Resist. 2024 Jul 4;17:2773-2783. doi: 10.2147/IDR.S455515. eCollection 2024. PMID 38979062
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2661041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants hospitalized for Community Acquired Pneumonia (CAP) or Complicated Soft Skin Tissue Infections (cSSTI) and treated with four or more consecutive intravenous (IV) doses of Zinforo (ceftaroline fosamil) in a usual care setting on or before 31-May-2019, were included. Data was collected retrospectively from hospital records and evaluated over approximately 14 months of this study.
Groups:
- Participants With CAP: Participants hospitalized for CAP and treated with 4 or more IV doses of Zinforo on or before 31-May-2019 were observed during this retrospective chart review study. The recommended dose of Zinforo was 600 milligram (mg) administered every 12 hours by intravenous infusion over 60 minutes for 5 to 7 days.
- Participants With cSSTI: Participants hospitalized for cSSTI and treated with 4 or more IV doses of Zinforo on or before 31-May-2019 were observed during this retrospective chart review study. The recommended dose of Zinforo was 600 mg administered every 12 hours by intravenous infusion over 60 minutes for 5 to 14 days.
Period: Overall Study
Arm/Group | Participants With CAP | Participants With cSSTI
Started | 185 | 132
Completed | 185 | 132
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants with the respective type of infection who were eligible for the study and whose data was entered into the study database.
Groups:
- Participants With CAP: Participants hospitalized for CAP and treated with 4 or more IV doses of Zinforo on or before 31-May-2019 were observed during this retrospective chart review study. The recommended dose of Zinforo was 600 mg administered every 12 hours by intravenous infusion over 60 minutes for 5 to 7 days.
- Total: Total of all reporting groups
Arm/Group | Participants With CAP | Participants With cSSTI | Total
Number analyzed (Participants) | 185 | 132 | 317
Age, Customized [Count of Participants; unit: Participants]
  18 to less than or equal to 65 years | 90 | 83 | 173
  Greater than 65 years | 95 | 49 | 144
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 55 | 131
  Male | 109 | 77 | 186
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response
Description: Clinical response in CAP was defined as participants demonstrating clinical stability (i.e., according to the Infectious Disease Society of America [IDSA] guidelines a temperature of less than or equal to (<=) 37.8 degree Celsius, heart rate of <=100 beats per minute, respiratory rate of <=24 breaths per minute, systolic blood pressure of greater than or equal to (>=) 90 millimeters of mercury (mmHg), oxygen saturation of >=90%, and confusion/disorientation recorded as absent) and clinical improvement (i.e., improvement of at least 1 of 4 symptoms present at Baseline [i.e., cough, dyspnea, pleuritic chest pain, sputum production] with worsening of none). Clinical response in cSSTI participants was defined as >=20% reduction from baseline infection area and cessation of spread measured by total infection area.
Time Frame: Day 1 of Zinforo treatment till end of Zinforo treatment: up to maximum of 35 days for CAP; up to maximum of 60 days for cSSTI (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 151 | 118

2. Primary Outcome: Time to Clinical Response
Description: Clinical response in CAP was defined as participants demonstrating clinical stability (i.e., according to the IDSA guidelines a temperature of <=37.8 degree Celsius, heart rate of <=100 beats per minute, respiratory rate of <=24 breaths per minute, systolic blood pressure of >=90 mmHg, oxygen saturation of >=90%, and confusion/disorientation recorded as absent) and clinical improvement (i.e., improvement of at least 1 of 4 symptoms present at Baseline (i.e., cough, dyspnea, pleuritic chest pain, sputum production) with worsening of none). Clinical response in cSSTI participants was defined as >=20% reduction from baseline infection area and cessation of spread measured by total infection area.
Time Frame: as for outcome 1
Population: Full analysis set included all participants with the respective type of infection who were eligible for the study and whose data was entered into the study database. Here, ''Overall number of participants analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 151 | 118
Days | 4 [0 to 18] | 4 [0 to 26]

3. Primary Outcome: Number of Participants Who Achieved Clinical Cure
Description: Clinical cure for both CAP and cSSTI was defined as the resolution of clinical features or improvement status requiring no further antibiotic therapy. Participants who achieved clinical cure were reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 115 | 72

4. Primary Outcome: Time to Clinical Cure
Description: Clinical cure for both CAP and cSSTI was defined as the resolution of clinical features or improvement status requiring no further antibiotic therapy. Time taken to achieve the clinical cure was reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 115 | 72
Days | 7 [1 to 25] | 5 [1 to 28]

5. Primary Outcome: Number of Participants With Clinical Failure
Description: Clinical failure for both CAP and cSSTI was defined as any of the following: treatment modification due to adverse event (AE); drug-drug interaction; insufficient response (followed by switch); death due to index infection; death due to other cause; relapse or recurrence.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 34 | 14

6. Primary Outcome: CAP: Number of Participants According to Reasons for Clinical Failure
Description: Clinical failure was defined as any of the following: treatment modification due to AE; drug-drug interaction; insufficient response (followed by switch); death due to index infection; death due to other cause; relapse or recurrence. Number of participants with CAP, according to the reasons for their clinical failure were reported in this outcome measure. Only those reasons which had at least 1 participant has been reported.
Time Frame: Day 1 of Zinforo treatment till end of Zinforo treatment, up to maximum of 35 days (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 34
Participants
  Insufficient response | 21
  Death due to index infection | 7
  Death due to other | 2
  Relapse or recurrence | 2
  Unknown | 2

7. Primary Outcome: cSSTI: Number of Participants According to Reasons for Clinical Failure
Description: Clinical failure was defined as any of the following: treatment modification due to AE; drug-drug interaction; insufficient response (followed by switch); death due to index infection; death due to other cause; relapse or recurrence. Number of participants with cSSTI, according to the reasons for their clinical failure were reported in this outcome measure. Only those reasons which had at least 1 participant has been reported.
Time Frame: Day 1 of Zinforo treatment till end of Zinforo treatment, up to maximum of 60 days (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 14
Participants
  Treatment modification due to AE | 1
  Insufficient response | 10
  Relapse or recurrence | 3

8. Primary Outcome: CAP Only: Time to Clinical Stability
Description: Clinical stability was defined according to the IDSA guidelines as temperature of <=37.8 degree Celsius, heart rate of <=100 beats per minute, respiratory rate of <=24 breaths per minute, systolic blood pressure of >=90 mmHg, oxygen saturation of >=90%, and confusion/disorientation recorded as absent. The time to achieve clinical stability was reported in this outcome measure.
Time Frame: as for outcome 6
Population: Full analysis set included all participants with the respective type of infection who were eligible for the study and whose data was entered into the study database. This outcome measure was planned to be analyzed only in CAP participants.
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Days | 3 [0 to 17]

9. Primary Outcome: CAP Only: Time to Clinical Improvement
Description: Clinical improvement was defined as improvement of at least 1 of 4 symptoms present at Baseline (i.e., cough, dyspnea, pleuritic chest pain, sputum production) with worsening of none. The time to clinical improvement was reported in this outcome measure.
Time Frame: Baseline (before Day 1 of Zinforo treatment) till end of Zinforo treatment, up to maximum of 35 days [from the retrospective data evaluated in approximately 14 months of the study]
Population: as for outcome 8
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Days | 3 [0 to 18]

10. Primary Outcome: CAP: Number of Participants With Early Response Within 4 Days
Description: Clinical response in CAP was defined as participants demonstrating clinical stability (i.e., according to the IDSA guidelines a temperature of <=37.8 degree Celsius, heart rate of <=100 beats per minute, respiratory rate of <=24 breaths per minute, systolic blood pressure of >=90 mmHg, oxygen saturation of >=90%, and confusion/disorientation recorded as absent) and clinical improvement (i.e., improvement of at least 1 of 4 symptoms present at Baseline [i.e., cough, dyspnea, pleuritic chest pain, sputum production] with worsening of none). Participants with CAP who showed response within 4 days after treatment with Zinforo were reported in this outcome measure.
Time Frame: Within 4 days after treatment with Zinforo (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants | 79

11. Primary Outcome: cSSTI: Number of Participants With Early Response Within 3 Days
Description: Clinical response in cSSTI participants was defined as >=20% reduction from baseline infection area and cessation of spread measured by total infection area. Participants with cSSTI who showed response within 3 days after treatment with Zinforo were reported in this outcome measure.
Time Frame: Within 3 days after treatment with Zinforo (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 132
Participants | 20

12. Primary Outcome: cSSTI Only: Time to Greater Than or Equal to (>=) 20% Reduction From Baseline in Infection Area
Description: The response to treatment in cSSTI participants was measured as >=20% reduction from baseline in infection area.
Time Frame: Baseline (before Day 1 of treatment) till end of treatment, up to maximum of 60 days [from the retrospective data evaluated in approximately 14 months of the study]
Population: Full analysis set included all participants with the respective type of infection who were eligible for the study and whose data was entered into the study database. This outcome measure was planned to be analyzed only in cSSTI participants. Here, ''Overall number of participants analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 118
Days | 3 [0 to 10]

13. Primary Outcome: cSSTI Only: Time to Cessation of Spread Measured by Total Infection Area
Description: The response to treatment in cSSTI participants was measured as cessation of spread of infection measured by total infection area.
Time Frame: as for outcome 7
Population: as for outcome 12
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 118
Days | 2 [0 to 26]

14. Primary Outcome: cSSTI Only: Time to Cessation of Spread Measured by Infection Length and Width
Description: Time taken for the cessation of spread of infection as measured by length and width of the infected area was reported in this outcome measure.
Time Frame: as for outcome 7
Population: as for outcome 12
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 118
Days | 2 [0 to 7]

15. Primary Outcome: Number of Participants According to Discharge Status
Description: Participants were categorized based on the discharge status in this outcome measure.
Time Frame: At discharge from hospital: any day till 102 days for CAP; any day till 162 days for cSSTI (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Died in the hospital | 18 | 6
  Discharged to a nursing home or extended care facility | 28 | 23
  Discharged to independent living (with or without support) | 138 | 101
  Other | 1 | 2

16. Primary Outcome: Number of Participants With Re-hospitalization Within 30 Days of Discharge
Description: The number of participants who were re-hospitalized within 30 days of discharge were reported in this outcome measure.
Time Frame: Within 30 days after discharge from hospital (discharge was any day till 102 days for CAP; any day till 162 days for cSSTI) [from the retrospective data evaluated in approximately 14 months of the study]
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 20 | 13

17. Primary Outcome: Number of Participants According to Vital Status Within 30 Days of Discharge
Description: The number of participants were classified according to the vital status in this outcome measure.
Time Frame: as for outcome 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Participant is still alive | 126 | 98
  Participant is deceased | 31 | 15
  Unknown | 28 | 19

18. Primary Outcome: Number of Participants According to Minimum Inhibitory Concentration (MIC) Assessment
Description: MIC was defined as the lowest concentration of an antimicrobial that will inhibit the visible growth of a microorganism. Participants were categorized as Yes, No or Unknown against being assessed for MIC.
Time Frame: From 1 week before Zinforo treatment through 24 hours post discontinuation of Zinforo treatment during index hospitalization (102 days for CAP; 162 days for cSSTI) [from retrospective data evaluated in approximately 14 months of study]
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Yes | 23 | 28
  No | 161 | 94
  Unknown | 1 | 10

19. Primary Outcome: Day of MIC Assessment Since Index Hospitalization
Description: Day of MIC assessment since the index hospitalization was reported in this outcome measure. Index hospitalization was first hospitalization on or before May 31, 2019 where Zinforo was administered for the treatment of CAP or cSSTI.
Time Frame: From Day 1 of Index hospitalization till MIC assessment, any day till 102 days for CAP; any day till 162 days for cSSTI (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 23 | 28
Days | 1 [0 to 10] | 4 [-10 to 47]

20. Primary Outcome: Number of Participants According to MIC of Antibacterial Drugs Assessed Based on Pathogens
Description: Pathogens for bacterial pneumonia were identified by blood, respiratory (e.g., sputum, bronchoalveolar lavage), or pleural effusion cultures and pathogens for cSSTI were identified blood or skin/soft tissue/bone/wound cultures. Number of participants with MIC of antibacterial drugs for pathogens isolated from samples were reported in this outcome measure.
Time Frame: as for outcome 18
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 23 | 28
Participants
  MIC of ceftaroline for all isolated pathogens | 5 | 7
  MIC of oxacillin, vancomycin, linezolid, and daptomycin for Staphylococcus aureus | 12 | 20
  MIC of ceftriaxone for Methicillin-Susceptible Staphylococcus aureus (MSSA) | 3 | 6
  MIC of penicillin and ceftriaxone for Streptococcus pneumonia | 10 | 0

21. Primary Outcome: Number of Participants With Serious Adverse Events
Description: An SAE was defined as any untoward medical occurrence at any dose that resulted in any of the following outcomes: death; life-threatening; hospitalization/prolongation of hospitalization; persistent/significant disability/incapacity; congenital anomaly/birth defect; or that was considered as an important medical event.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 0 | 2

22. Primary Outcome: Number of Participants With Medical Conditions Presented at Index Hospitalization
Description: The number of participants who had any medical conditions at the time of index hospitalization were reported in this outcome measure. Medical conditions that were considered included Human Immunodeficiency Virus (HIV) infection, alcohol abuse, cancer/malignancy, cerebrovascular disease, chronic dialysis within the past 30 days, chronic obstructive pulmonary disease, chronic renal disease, congestive heart failure, decompensated cirrhosis, diabetes mellitus, immunosuppressive disease, influenza, injection drug use, end stage liver disease, peripheral vascular disease, respiratory disease or any other relevant condition(s) or disease(s) that required chronic drug treatment. Index hospitalization was first hospitalization on or before May 31, 2019 where Zinforo was administered for the treatment of CAP or cSSTI.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 147 | 99

23. Primary Outcome: Number of Participants With Hospitalization for Any Reason in the 3 Months Before the Index Hospitalization
Description: The number of participants who had hospitalization for any reason, 3 months before the index hospitalization were reported in this outcome measure. Index hospitalization was first hospitalization on or before May 31, 2019 where Zinforo was administered for the treatment of CAP or cSSTI.
Time Frame: 3 months prior to index hospitalization (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 34 | 44

24. Primary Outcome: Number of Participants With Invasive Major Surgical Treatment in the 3 Months Before the Index Hospitalization
Description: The number of participants who had undergone surgical treatments, 3 months before to the index hospitalization were reported in this outcome measure.
Time Frame: 3 months prior to index hospitalization (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 5 | 24

25. Primary Outcome: Number of Participants According to Therapies Received in the 3 Months Before the Index Hospitalization
Description: Number of participants according to therapies received in the 3 months prior to index hospitalization were reported in this outcome measure. One participant could receive more than one therapy.
Time Frame: 3 months prior to index hospitalization (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Antimicrobial (e.g. antibiotics, antivirals) | 47 | 56
  Immunosuppressors/ immunomodulators | 21 | 19
  Anticoagulants | 38 | 45
  Non-steroid anti-inflammatory agents (NSAIs) | 13 | 25
  Home infusion therapy | 3 | 2
  Home wound care provided by a medical professional | 6 | 5
  None | 103 | 39

26. Primary Outcome: Number of Participants With Radiographic Findings in Tests for CAP
Description: Participants were categorized according to radiographic findings in the tests conducted for diagnosis of CAP infection in this outcome measure. One participant could have more than one radiographic finding.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants
  Infiltrate | 130
  Consolidation | 68
  Pleural effusion | 48
  Other findings | 30
  None of the above | 3

27. Primary Outcome: CAP: Number of Participants With Triggering Signs and Symptoms at Index Hospitalization
Description: Participants were categorized according to triggering signs and symptoms at CAP diagnosis and recorded at index hospital admission were reported in this outcome measure. The observed signs and symptoms were dyspnea, tachypnea, or hypoxemia (oxygen [O2] saturation < 90% on room air or partial pressure of oxygen (pO2) < 60 mmHg), Fever (>38 degree Celsius[C]oral; > 38.5 degree C rectally or tympanically) or hypothermia (< 35 degree C), White Blood Cell (WBC) count > 10,000 cells/cubic millimeter(mm³) or < 4,500 cells/mm³. One participant could have more than one signs or symptoms.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants
  New or increased cough | 129
  Purulent sputum or change in sputum character | 80
  Auscultatory findings consistent with pneumonia | 138
  Dyspnea, tachypnea, or hypoxemia (O2 saturation < 90% on room air or pO2 < 60 mmHg) | 148
  Fever (>38 degree C oral; > 38.5 degree C rectally or tympanically) or hypothermia (< 35 degree C) | 127
  WBC count > 10,000 cells/mm³ or < 4,500 cells/mm³ | 122

28. Primary Outcome: Number of Participants With Severe CAP
Description: Number of participants diagnosed with severe CAP were reported in this outcome measure.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants | 128

29. Primary Outcome: Number of Participants According to Type of Prognostic Scoring System Used to Assess CAP Severity
Description: In this outcome measure participants were categorized according to type of assessment used to assess CAP severity. Pneumonia severity index (PSI)/PORT score was used to calculate the probability of morbidity and mortality among participants with CAP. The score was used to predict the need for hospitalization in people with pneumonia. CURB- 65 was used to measure the confusion, blood urea, respiratory rate, blood pressure for the participants aged greater than or equal to 65 years. Multiple criteria to assess the severity of CAP exist. In this study severity was first globally assessed asking if a (any) criterion for severity of CAP would apply. In subsequent questions the details on the exact methods of the severity assessment were then asked. This included the information about PORT score / PSI, CURB-65 and recurrency of CAP.
Time Frame: At index hospitalization admission(from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants
  PORT Score / Pneumonia Severity Index | 18
  CURB-65 | 41
  Other | 15
  None | 71
  Unknown | 40

30. Primary Outcome: Time of CAP Diagnosis at Index Hospitalization
Description: The time taken (in days) taken to diagnose CAP in the participants prior to index hospitalization were reported in this outcome measure and this data was recorded at index hospitalization admission.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: Full analysis set included all participants with the respective type of infection who were eligible for the study and whose data was entered into the study database. This outcome measure was planned to be analyzed only in CAP participants. Here, ''Overall number of participants analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP
Number analyzed (Participants) | 99
Days | 1 [0 to 20]

31. Primary Outcome: Number of Participants With Recurrent CAP Infections at Index Hospitalization
Description: The number of participants with recurrent CAP infections were reported in this outcome measure.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants | 10

32. Primary Outcome: Number of Participants According to Microbiological CAP Diagnosis at Index Hospitalization
Description: The number of participants were classified according to the various pathogens identified during CAP diagnosis in this outcome measure.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants
  Streptococcus pneumonia | 44
  Escherichia coli | 2
  Hemophilus influenza | 3
  H. Parainfluenza | 1
  Legionella spp. | 2
  Staphylococcus aureus | 4
  Methicillin resistance Staphylococcus aureus | 14
  Methicillin susceptible Staphylococcus. aureus | 15
  Klebsiella pneumonia | 3
  Other enterobacteria | 2
  Pseudomonas aeruginosa | 1
  Other microorganism | 26
  Unknown | 15
  None of the above | 72

33. Primary Outcome: Number of Participants According to Type of Investigation Performed for Positive Microbiological CAP Diagnosis at Index Hospitalization
Description: The number of participants were classified according to the type of investigations performed for the microbiological CAP diagnosis and were reported in this outcome measure.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: Analysis population included all eligible participants whose data were retrieved from hospital medical records and assessed. This outcome measure was planned to be analyzed only in CAP participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants
  Sputum examination | 33
  Blood culture | 39
  Bronchoalveolar lavage or bronchial brush examination | 10
  Pleural fluid sample examination | 4
  Legionella antigen test in urine | 5
  Pneumococcal antigen test in urine | 30
  Other | 17

34. Primary Outcome: CAP: Number of Participants With Polymerase Chain Reaction (PCR) Determination of H1N1 Influenza Virus at Index Hospitalization
Description: In this outcome measure number of participants who had H1N1 Influenza virus determined using PCR were reported.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants | 71

35. Primary Outcome: CAP: Number of Participants According to Influenza Vaccination Status During 12 Months Prior to Index Hospitalization
Description: The number of participants according to the status of influenza vaccination were reported in this outcome measure, as vaccinated: Yes, No and Unknown.
Time Frame: 12 months prior to index hospitalization (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants
  Yes | 32
  No | 64
  Unknown | 89

36. Primary Outcome: CAP: Number of Participants According to Pneumococcal Vaccination Status at Index Hospitalization
Description: The number of participants according to the status of pneumococcal vaccination were reported in this outcome measure.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants
  Yes | 18
  No | 76
  Unknown | 91

37. Primary Outcome: CAP: Number of Participants According to the Biomarkers Used for Monitoring Clinical Evolution at Index Hospitalization
Description: The number of participants were classified according to the biomarkers used for monitoring the state of CAP in this outcome measure.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP
Number analyzed (Participants) | 185
Participants
  C-reactive protein (CRP) | 182
  Procalcitonin | 73
  Other biomarker | 8
  None of the above | 2

38. Primary Outcome: cSSTI: Number of Participants According to Type of Lesions Involved at Index Hospitalization
Description: The number of participants classified according to the types of lesions involved in the cSSTI infection were reported in this outcome measure. One participant could have more than one type of lesion.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: Full analysis set included all participants with the respective type of infection who were eligible for the study and whose data was entered into the study database. This outcome measure was planned to be analyzed only in cSSTI participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 132
Participants
  Abscess | 45
  Cellulitis/fasciitis | 82
  Post-traumatic wound | 9
  Post-surgical wound | 26
  Decubitus ulcer | 5
  Diabetic leg ulcer | 5
  Peripheral vascular disease ulcer | 3
  Bite | 1
  Unknown | 1
  None of the above | 2

39. Primary Outcome: cSSTI: Number of Participants According to Type of Body Area Involved at Index Hospitalization
Description: The number of participants were classified according to the body area involved in cSSTI are reported in this outcome measure. One participant could have more than one type of body area involvement.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 132
Participants
  Head | 13
  Hand | 3
  Upper extremities | 14
  Lower extremities | 74
  Thorax | 19
  Abdomen | 14
  Genitalia | 9
  Unknown | 1

40. Primary Outcome: cSSTI: Number of Participants According to Area of Extension of Skin Infection at Index Hospitalization
Description: The number of participants were classified according to the extent of skin that was affected with the infection in this outcome measure.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 132
Participants
  Less than (<) 5 centimeter square (cm^2) | 12
  5-10 cm^2 | 31
  10-50 cm^2 | 34
  Greater than (>) 50 cm^2 | 8
  Unknown | 47

41. Primary Outcome: cSSTI: Number of Participants According to Level of Infections at Index Hospitalization
Description: The number of participants were classified according to the level of infections in this outcome measure.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 132
Participants
  Superficial | 51
  Deep incisional | 51
  Organ or space infection | 20
  Unknown | 10

42. Primary Outcome: cSSTI: Number of Participants According to Type of Anatomical Structures Affected at Index Hospitalization
Description: The number of participants were classified according to the anatomical structures involved in the infections in this outcome measure.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 132
Participants
  Epithelium | 61
  Epidermis | 92
  Dermis | 88
  Subcutaneous fat | 61
  Fascia | 23
  Muscle | 25
  Unknown | 23

43. Primary Outcome: Time of cSSTI Diagnosis at Index Hospitalization
Description: The time taken (in days) taken to diagnose cSSTI in the participants prior to index hospitalization were reported in this outcome measure and this data was recorded at index hospitalization admission.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 12
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 51
Days | 5 [0 to 100]

44. Primary Outcome: cSSTI: Number of Participants With Recurrent Infection at Index Hospitalization
Description: The number of participants that had recurrent cSSTI infections were reported in this outcome measure.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 132
Participants | 33

45. Primary Outcome: cSSTI: Number of Participants With Triggering Signs and Symptoms at Index Hospitalization
Description: The number of participants with triggering signs and symptoms during the cSSTI diagnosis were reported in this outcome measure. One participant could have more than one triggering signs and symptoms.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 132
Participants
  Purulent or seropurulent drainage/discharge | 65
  Bullae | 5
  Erythema | 106
  Fluctuance | 30
  Heat/localized warmth | 90
  Pain/tenderness to palpitation | 100
  Swelling/induration | 78
  Skin necrosis | 9
  Anesthesia | 1
  Crackling | 3
  Induration beyond the erythematous area | 17

46. Primary Outcome: Number of Participants According to Systemic Signs of cSSTI at Index Hospitalization
Description: The number of participants were classified according to the systemic signs observed Including temperature greater than (>) 30 degree Celsius, White blood cell count >10,000 cells per millimeter cube(/mm3) or <4,500/mm3 or immature neutrophils >10%, septic shock, organ dysfunction and none of the above mentioned were reported. One participant could have more than one systemic sign.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 132
Participants
  Temperature > 38 degree Celsius | 77
  White blood cell count | 108
  Septic shock | 4
  Organ dysfunction | 13
  None of the above | 1

47. Primary Outcome: cSSTI: Number of Participants According to Type of Diagnostic Tests Conducted at Index Hospitalization
Description: The number of participants classified according to the diagnostic tests conducted to diagnose cSSTI were reported in this outcome measure. One participant could have more than one type of diagnostic test.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 132
Participants
  Blood cultures | 85
  Superficial swab and culture | 40
  Needle aspiration | 14
  Skin biopsy | 7
  Surgical sample | 22
  X-ray | 31
  Ultrasound | 58
  Computed Tomography (CT)/ Magnetic Resonance Imaging (MRI) | 35
  Unknown/not performed | 6

48. Primary Outcome: cSSTI: Number of Participants According to Microbiologic Diagnosis at Index Hospitalization
Description: Pathogens identified by blood or skin/soft tissue/bone/wound cultures were recorded for participants with cSSTI.
Time Frame: At index hospitalization admission (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With cSSTI
Number analyzed (Participants) | 132
Participants
  Methicillin resistance Staphylococcus aureus | 24
  Methicillin susceptible S. aureus (MSSA) | 23
  Staphylococcus coagulase negative | 8
  Streptococcus pneumonia | 1
  Streptococcus pyogenes | 4
  Streptococcus agalactiae | 1
  Enterococcus faecalis | 2
  Gram-negative bacilli | 12
  Non-fermenting enterobacteria | 1
  Other strict anaerobic bacteria | 1
  Other microorganism | 8
  Mixed flora | 1
  Unknown | 24
  None of the above | 40

49. Primary Outcome: Number of Participants According to Class of Antibiotics Received Prior to Zinforo Treatment During Index Hospitalization
Description: The number of participants were classified according to types of antibiotics that they received prior to Zinforo and reported in this outcome measure.
Time Frame: Before Zinforo treatment initiation during index hospitalization, index hospitalization was of 102 days for CAP; 162 days for cSSTI (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 134 | 87
Participants
  Aminoglycoside | 5 | 6
  Betalactam | 17 | 20
  Carbapenem | 12 | 4
  Ceftriaxone | 45 | 10
  Cephalosporins | 19 | 16
  Glycopeptide | 4 | 18
  Macrolide | 13 | 23
  Betalactam/Combination | 36 | 6
  Quinolone | 50 | 21
  Sulfonamide | 37 | 10
  Clindamycin | 1 | 4
  Other antibiotic agent | 15 | 8
  Unknown | 17 | 31

50. Primary Outcome: Number of Participants According to Lines of Pre-Zinforo Therapies During Index Hospitalization
Description: The number of participants were classified according to the lines of therapy in this outcome measure.
Time Frame: as for outcome 49
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 134 | 87
Participants
  First | 134 | 87
  Second | 85 | 58
  Third | 40 | 24
  Fourth | 20 | 13
  Fifth | 5 | 5
  Sixth | 2 | 3
  Seventh | 1 | 3
  Eighth | 1 | 3
  Nineth | 0 | 1
  Tenth | 0 | 1

51. Primary Outcome: Number of Participants According to Routes of Administration for Pre-Zinforo Treatment During Index Hospitalization
Description: The number of participants were classified according to various routes of administration for pre-Zinforo treatment and were reported in this outcome measure.
Time Frame: as for outcome 49
Population: Full analysis set included all participants with the respective type of infection who were eligible for the study and whose data was entered into the study database. Here, ''Overall number of participants'' analyzed signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 134 | 87
Participants
  Oral | 44 | 31
  Intra-venous | 111 | 73
  Intra-muscular | 7 | 0
  Subcutaneous | 0 | 1
  Unknown | 4 | 3

52. Primary Outcome: Duration of Pre-Zinforo Treatment During Index Hospitalization
Time Frame: as for outcome 49
Population: as for outcome 51
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 134 | 87
Days | 6 [0 to 45] | 8 [1 to 40]

53. Primary Outcome: Time From Symptom Onset to First Dose of Pre-Zinforo Treatment
Time Frame: as for outcome 49
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 134 | 87
Days | 3 [0 to 20] | 2 [0 to 30]

54. Primary Outcome: Number of Participants According to Types of Pre-Zinforo Treatment During Index Hospitalization
Description: The number of participants were classified according to types of Pre-Zinforo treatment and were reported in this outcome measure. One participant could have more than one type of pre-Zinforo treatment.
Time Frame: as for outcome 49
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 134 | 87
Participants
  Empiric | 129 | 74
  Definitive/Specific | 13 | 19
  Unknown | 6 | 10

55. Primary Outcome: Number of Doses Administered for Pre-Zinforo Treatment During Index Hopsitalization
Time Frame: as for outcome 49
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 134 | 87
Doses | 2.02 (0.93) | 2.18 (1.54)

56. Primary Outcome: Number of Participants With Pre-Zinforo Treatment Modification During Index Hospitalization
Description: The number of participants who had pre-Zinforo treatment modification were reported in this outcome measure.
Time Frame: as for outcome 49
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 134 | 87
Participants | 91 | 60

57. Primary Outcome: Number of Participants According to Reasons for Pre-Zinforo Treatment Modification
Description: The number of participants classified according to the reasons for pre-Zinforo treatment modification were reported in this outcome measure. One participant could have more than one reason for treatment modification. Index hospitalization was first hospitalization on or before May 31, 2019 where Zinforo was administered for the treatment of CAP or cSSTI. One participant could have more than one reason for treatment modification.
Time Frame: as for outcome 49
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 91 | 60
Participants
  Adverse event | 5 | 3
  Insufficient response | 58 | 42
  Possible interaction with other drug | 1 | 1
  Streamlining | 29 | 9
  Other | 14 | 16

58. Primary Outcome: Number of Participants Based on Treatment Response to Pre-Zinforo Treatment During Index Hospitalization
Description: Treatment response was defined according to the following criteria: CAP participants who demonstrated clinical stability (defined according to the Infectious Diseases Society of America [IDSA] guidelines as temperature of ≤37.8 C°, heart rate of ≤100 beats/min, respiratory rate of ≤24 breaths/min, systolic blood pressure of ≥90mmHg, oxygen saturation of ≥90%, and confusion/disorientation recorded as absent) and clinical improvement{defined as improvement of at least 1 of 4 symptoms present at baseline (i.e., cough, dyspnea, pleuritic chest pain, sputum production) with worsening of none}. cSSTI participants: ≥20% reduction from baseline infection area and cessation of spread measured by total infection area. The number of participants were classified according to treatment response to pre-Zinforo treatment and were reported in this outcome measure.
Time Frame: as for outcome 49
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 134 | 87
Participants
  Response | 12 | 17
  No response | 89 | 14
  Unknown | 33 | 62

59. Primary Outcome: Time to Treatment Modification From Initial Dose of Pre-Zinforo Treatment
Description: The time (days) taken for modification from initial dose of pre-Zinforo treatment were reported in this outcome measure.
Time Frame: Before Zinforo treatment initiation during index hospitalization, index hospitalization was maximum of 102 days for CAP; maximum of 162 days for cSSTI (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 91 | 60
Days | 2 [0 to 13] | 3 [0 to 20]

60. Primary Outcome: Number of Participants With Insufficient Response to Pre-Zinforo Treatment During Index Hospitalization
Description: The number of participants with insufficient response to pre-Zinforo treatment were reported in this outcome measure.
Time Frame: as for outcome 59
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 134 | 87
Participants | 58 | 42

61. Primary Outcome: Duration of Zinforo Treatment During Index Hospitalization
Description: The duration of Zinforo treatment for CAP and cSSTI infections were reported in this outcome measure.
Time Frame: Day 1 of Zinforo treatment till end of Zinforo treatment, during index hospitalization, index hospitalization was maximum of 102 days for CAP; maximum of 162 days for cSSTI (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Days | 7 [2 to 35] | 8 [2 to 60]

62. Primary Outcome: Time From Admission to First Dose of Zinforo During Index Hospitalization
Description: The time taken from admission to the administration of first dose of Zinforo was reported in this outcome measure.
Time Frame: as for outcome 61
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Days | 1 [0 to 36] | 1 [0 to 60]

63. Primary Outcome: Time From Symptom Onset to First Dose of Zinforo During Index Hospitalization
Description: The time taken for the symptom onset to the administration of first dose of Zinforo was reported in this outcome measure.
Time Frame: During index hospitalization, index hospitalization was maximum of 102 days for CAP; maximum of 162 days for cSSTI (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Days | 6 [0 to 38] | 7 [0 to 64]

64. Primary Outcome: Number of Participants According to Types of Treatment for Zinforo
Description: The number of participants classified according to the types of treatment for Zinforo were reported in this outcome measure. Types included empiric, definitive/specific and unknown. Empiric was defined as therapy administered to participants prior to the results of blood culture and susceptibility tests. Definitive was defined as therapy administered after the test results were received.
Time Frame: as for outcome 63
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Empiric | 138 | 84
  Definitive/Specific | 41 | 43
  Unknown | 6 | 5

65. Primary Outcome: Daily Dose of Zinforo
Time Frame: as for outcome 61
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Milligrams | 1183.24 (412.69) | 1239.39 (402.43)

66. Primary Outcome: Number of Infusions Administered Daily for Zinforo
Time Frame: as for outcome 61
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Infusions
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Infusions | 2.28 (0.47) | 2.27 (0.46)

67. Primary Outcome: Number of Participants According to Locations of Zinforo Administration
Description: The number of participants were classified according to the locations where Zinforo was administered were reported in this outcome measure. One participant could have more than one location of Zinforo administration.
Time Frame: as for outcome 61
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Intensive Care Unit (ICU) | 66 | 11
  General ward | 115 | 114
  At home | 1 | 14
  Medical clinic | 30 | 14
  Out-patient setting | 0 | 2

68. Primary Outcome: Number of Participants Administered Zinforo as Monotherapy or Combination Therapy
Description: The number of participants were classified according to Zinforo administration as monotherapy or combination therapy were reported in this outcome measure.
Time Frame: as for outcome 61
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Monotherapy | 56 | 78
  Combination therapy | 129 | 54

69. Primary Outcome: Number of Participants Receiving Concomitant Therapies Along With Zinforo
Description: Number of participants who received concomitant therapies along with Zinforo were reported in this outcome measure.
Time Frame: as for outcome 61
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 131 | 92

70. Primary Outcome: Number of Participants According to Type of Antibiotics Received for Index Infection After Zinforo Treatment
Description: The number of participants were classified according to types of antibiotics received for index infection (CAP and cSSTI) after the Zinforo treatment were reported in this outcome measure. One participant could receive more than one type of antibiotic.
Time Frame: Post Zinforo treatment, during index hospitalization, index hospitalization was maximum of 102 days for CAP; maximum of 162 days for cSSTI (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 99 | 75
Participants
  Aminoglycoside | 9 | 3
  Betalactam | 13 | 4
  Carbapenem | 8 | 5
  Ceftriaxone | 18 | 15
  Glycopeptide | 7 | 5
  Macrolide | 12 | 2
  Betalactam/Combination | 27 | 12
  Quinolone | 45 | 28
  Sulfonamide | 12 | 2
  Clindamycin | 32 | 21
  Other antibiotic agent | 12 | 20
  Linezolid | 0 | 2
  Unknown | 9 | 0

71. Primary Outcome: Number of Participants According to Lines of Therapy for Post-Zinforo Treatment
Description: The number of participants were classified according to the lines of therapy for post-Zinforo treatment were reported in this outcome measure.
Time Frame: as for outcome 70
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 99 | 75
Participants
  First | 1 | 2
  Second | 45 | 46
  Third | 40 | 20
  Fourth | 51 | 21
  Fifth | 26 | 11
  Sixth | 25 | 5
  Seventh | 5 | 5
  Eighth | 8 | 2
  Nineth | 3 | 4
  Tenth | 0 | 1
  Eleventh | 0 | 1
  Twelfth | 0 | 1

72. Primary Outcome: Number of Participants According to Route of Administration for Post-Zinforo Treatment
Description: The number of participants were classified according to routes of administration for post-Zinforo treatment were reported in this outcome measure.
Time Frame: CAP (up to maximum of 102 days), cSSTI (up to maximum of 162 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Oral | 92 | 81
  Intra-venous | 112 | 38

73. Primary Outcome: Duration From Zinforo Discontinuation to Initiation of New Treatment
Description: The duration in days from Zinforo treatment discontinuation to initiation of new treatment were reported in this outcome measure.
Time Frame: as for outcome 70
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Days | 1 [0 to 56] | 1 [0 to 36]

74. Primary Outcome: Number of Doses Administered for Post Zinforo Treatment
Time Frame: as for outcome 70
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Doses | 11.05 (14.82) | 16.38 (21.81)

75. Primary Outcome: Number of Participants According to Reasons for Switching to Post-Zinforo Treatment
Description: The number of participants were classified according to the reasons for switching to post-Zinforo treatment were reported in this outcome measure. One participant could have more than one reason for switch.
Time Frame: as for outcome 70
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Lack of efficacy of previous treatment | 39 | 9
  Side effect of previous treatment | 1 | 9
  Results of susceptibility test/pathogen identification | 26 | 14
  Other | 124 | 81
  Unknown | 14 | 6

76. Primary Outcome: Number of Participants Based on Treatment Response to Post-Zinforo Treatment
Description: Clinical response in CAP:participants demonstrating clinical stability(i.e.,according to IDSA guidelines:temperature of<=37.8 degree Celsius,heart rate of <=100 beats per minute,respiratory rate of <=24 breaths per minute,systolic blood pressure of >=90 mmHg,oxygen saturation of >=90%,confusion/disorientation recorded as absent),clinical improvement(i.e.,improvement of at least 1 of 4 symptoms present at Baseline(i.e.,cough,dyspnea,pleuritic chest pain,sputum production)with worsening of none).Clinical response in cSSTI participants:>=20% reduction from baseline infection area,cessation of spread measured by total infection area.Clinical failure for both CAP and cSSTI:any of the following:treatment modification due to AE;drug-drug interaction;insufficient response(followed by switch);death due to index infection;death due to other cause;relapse or recurrence. Number of participants classified according to treatment responses to post-Zinforo treatment reported in this outcome measure.
Time Frame: as for outcome 70
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Clinical response | 155 | 95
  Clinical failure | 26 | 4
  Unknown | 23 | 20

77. Primary Outcome: Number of Participant According to Type of Location for Post-Zinforo Treatment Administration
Description: The number of participants were classified according to the locations in which post-Zinforo treatment was administered. One participant could have more than one location of administration.
Time Frame: as for outcome 70
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  ICU | 70 | 1
  General ward | 86 | 42
  At home | 64 | 70
  Out-patient setting | 9 | 16
  Medical clinic | 6 | 5
  Other | 0 | 1

78. Primary Outcome: Number of Participants Who Achieved Clinical Response to Post-Zinforo Treatment
Description: as for outcome 2
Time Frame: as for outcome 70
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 139 | 89

79. Primary Outcome: Number of Participants According to Reasons for Clinical Failure to Post-Zinforo Treatment
Description: Clinical failure for both CAP and cSSTI was defined as any of the following: treatment modification due to AE; drug-drug interaction; insufficient response (followed by switch); death due to index infection; death due to other cause; relapse or recurrence. The number of participants were classified according to the reasons for clinical failure post-Zinforo treatment were reported in this outcome measure.
Time Frame: as for outcome 70
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 26 | 4
Participants
  Treatment modification due to adverse event | 2 | 0
  Insufficient response | 14 | 1
  Relapse/reoccurrence | 1 | 0
  Death due to infection | 6 | 0
  Death due to other | 3 | 3

80. Primary Outcome: Duration of Index Hospitalization
Description: Index hospitalization was first hospitalization on or before May 31, 2019 where Zinforo was administered for the treatment of CAP or cSSTI.
Time Frame: Day 1 of admission of index hospitalization to discharge from hospital (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Days | 12 [3 to 102] | 11 [3 to 162]

81. Primary Outcome: Duration in Intensive Care Unit
Time Frame: as for outcome 63
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Days | 0 [0 to 46] | 0 [0 to 41]

82. Primary Outcome: Number of Participants Who Received Renal Replacement Therapy Post Initiating Treatment With Zinforo
Description: The number of participants who received renal replacement therapy after initiating treatment with Zinforo were reported in this outcome measure.
Time Frame: Post initiation of Zinforo treatment, during index hospitalization, index hospitalization was maximum of 102 days for CAP; maximum of 162 days for cSSTI (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 5 | 2

83. Primary Outcome: Number of Participants According to Treatments Received During Index Hospitalization
Description: The number of participants were classified according to treatments received during index hospitalization were reported in this outcome measure.
Time Frame: as for outcome 63
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Surgery related to the infection | 5 | 37
  Surgery unrelated to the infection | 1 | 0
  Blood pressure support | 44 | 12
  Blood pressure support: Fluid resuscitation | 32 | 7
  Blood pressure support: Vasopressors | 44 | 10
  Blood pressure support: Invasive procedures | 2 | 0
  None of the above | 139 | 90

84. Primary Outcome: Number of Participants Who Received Home-Based Care Through a Healthcare Agency
Description: The number of participants who received home-based care through a healthcare agency were reported in this outcome measure.
Time Frame: Within 30 days post discharge from index hospitalization (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 16 | 35

85. Primary Outcome: Number of Participants With Re-hospitalizations
Description: The number of participants who had re-hospitalizations were reported in this outcome measure.
Time Frame: as for outcome 84
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 20 | 13

86. Primary Outcome: Duration of Re-hospitalizations
Description: In this outcome measure, data is recorded for duration (in days) of re-hospitalization (if any) that happened within 30 days post discharge from index hospitalization.
Time Frame: Day 1 of re-hospitalization till discharge (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 20 | 13
Days | 10.5 [1 to 39] | 9 [2 to 30]

87. Primary Outcome: Number of Participants According to Reasons for Re-hozpitalization
Description: The number of participants were classified according to reasons for re-hospitalizations were reported in this outcome measure. Re-hospitalization (if any) that happened within 30 days post discharge from index hospitalization.
Time Frame: as for outcome 86
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 20 | 13
Participants
  For index infection | 7 | 3
  For other reason | 13 | 10

88. Primary Outcome: Number of Participants With Development of Sepsis During Index Hospitalization
Description: The number of participants who developed sepsis during index hospitalization were reported in this outcome measure.
Time Frame: as for outcome 63
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 38 | 29

89. Primary Outcome: Number of Participants With Quick Sepsis-Related Organ Failure Assessment (qSOFA) Conducted
Description: The qSOFA (also known as quickSOFA) was a bedside prompt that identified participants with suspected infection who are at greater risk for a poor outcome outside the intensive care unit (ICU). It used three criteria, assigning one point for low blood pressure Systolic blood pressure less than or equal to 100 millimeters of mercury (SBP<=100 mmHg), high respiratory rate greater than or equal to (>=) 22 breaths per min, or altered mentation (Glasgow coma scale<15).
Time Frame: as for outcome 63
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 74 | 40

90. Primary Outcome: Number of Participants Requiring Isolation
Description: The number of participants who required isolation were reported in this outcome measure.
Time Frame: as for outcome 63
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 20 | 10

91. Primary Outcome: Number of Participants Who Received Mechanical Ventilation, Oxygen Therapy and Parenteral Nutrition
Time Frame: as for outcome 63
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants
  Mechanical Ventilation | 56 | 11
  Oxygen Therapy | 37 | 6
  Parenteral Nutrition | 17 | 5

92. Primary Outcome: Number of Participants Who Suffered Acute Renal Failure Necessitating Renal Replacement
Description: The number of participants who suffered from acute renal failure and necessitated renal replacement were reported in this outcome measure.
Time Frame: as for outcome 63
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Participants | 11 | 4

93. Primary Outcome: Total Number of Doses of Zinforo Administered
Time Frame: as for outcome 61
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Doses | 18.96 (11.05) | 23.29 (18.2)

94. Primary Outcome: Total Number of Doses of Other Antibiotics Administered in Combination With Zinforo
Time Frame: as for outcome 61
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Doses | 8.48 (9.81) | 8.48 (9.81)

95. Primary Outcome: Total Dose of Other Antibiotics Administered Post Zinforo Treatment
Time Frame: as for outcome 70
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
Milligrams | 11.05 (14.82) | 11.05 (14.82)

96. Primary Outcome: Cost of Hospitalization
Description: The cost of hospitalization of standard level hospitals was calculated as total hospital cost= total number of bed days * per diem rate standard hospital general ward and the cost of hospitalization of advanced level hospitals was calculated as total number of bed days * per diem rate advanced hospital.
Time Frame: Day 1 of index hospitalization till discharge, index hospitalization was maximum of 102 days for CAP; maximum of 162 days for cSSTI (from the retrospective data evaluated in approximately 14 months of the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Participants With CAP | Participants With cSSTI
Number analyzed (Participants) | 185 | 132
US dollars
  Standard hospital cost | 9204.62 (12895.23) | 5196.2 (9070.35)
  Advanced level cost | 25408.01 (31704.58) | 20257.18 (36809.71)

ADVERSE EVENTS:
Time Frame: For adverse events: Day 1 of Zinforo treatment till end of Zinforo treatment: up to maximum of 35 days for CAP; up to maximum of 60 days for cSSTI; For death: Day 1 of index hospitalization up to 30 days of discharge, index hospitalization was maximum of 102 days for CAP; maximum of 162 days for cSSTI (from the retrospective data evaluated in approximately 14 months of the study)
Description: The adverse events attributed only to Zinforo treatment during index hospitalization as observed from medical records of participants were reported. There was no specific medical dictionary utilized to record adverse events.
Arm/Group | Participants With CAP | Participants With cSSTI
All-Cause Mortality (participants affected / at risk) | 31/185 | 15/132
Serious Adverse Events (participants affected / at risk) | 0/185 | 2/132
Other Adverse Events (participants affected / at risk) | 0/185 | 0/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With CAP (N=185) | Participants With cSSTI (N=132)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Drug hypersensitivity (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT04198571/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT04198571/SAP_001.pdf